CLINICAL TRIAL: NCT02273128
Title: Calcitonin Receptor Gene Polymorphisms in Patients With Osteoporosis and Chronic Periodontitis-An Observational Study
Brief Title: A Study to Assess the Disturbances in Calcitonin Gene in Patients With Gum Disease and Osteoporosis
Acronym: CTROP
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr,Anuradha Ankam, Post Graduate, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: D129206005
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Generalized Chronic Periodontitis; Osteoporosis
Keywords: Osteoporosis; Chronic Periodontitis; Calcitonin gene Polymorphism
MeSH Terms: conditions — Osteoporosis; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 2ml of blood sample from each subject was collected in EDTA containing vials and kept at -20 degrees until DNA extraction. The genomic DNA was isolated and C/T polymorphism in CTR gene was identified by PCR followed by restriction digestion pattern by Alu 1 restriction enzyme.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CTR Gene in Osteoporosis and Periodontitis: Patients aged between 35 - 60 yrs with Osteoporosis (BMD>-2.5) and Chronic Periodontitis (>3mm Pocket Probing Depth)
  Interventions: Genetic: CTR Gene

INTERVENTIONS:
Genetic: CTR Gene — 2ml blood sample collected from patients to extract DNA for Assessment of CTR Gene polymorphism
  Other Names: Calcitonin Gene, Hypocalcaemic agent

SUMMARY:
Osteoporosis and Periodontitis are multifactorial diseases which share common risk factors.The aim of the present study is to ellucidate polymorphisms in Calcitonin receptor gene? in patients with Osteoporosis and Periodontitis.

DETAILED DESCRIPTION:
Periodontitis is a polymicrobial inflammatory disease which includes various modifiable and nonmodifiable risk factors. The non modifiable risk factors include genetic polymorphisms like metabolism associated genetic polymorphisms ( Vitamin D and Calcitonin).

Osteoporosis is a systemic skeletal disease characterized by low bone mass and micro-architectural deterioration of bone tissue with consequent increase in bone fragility and susceptibility to fractures.

Bone loss is a common feature shared between periodontal disease and osteoporosis.

Out of all genetic factors Calcitonin gene polymorphism contributes to the development of both osteoporosis and chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Patients aged between 35.00 Year(s) to 60.00 Year(s) diagnosed with Osteoporosis and Chronic Periodontitis who are willing to participate in the study

Exclusion Criteria:

* Patients who are Systemically compromised and under medications such as steroids.
* Patients who smoke.Pregnant and lactating mothers are excluded from the study

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients both male and female aged between 35-60 Years with Osteoporosis and Chronic Periodontitis.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Calcitonin gene polymorphism | 5 Months
  Collection of blood samples and running the samples by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Anuradha Ankam, PG(Perio), Principal Investigator — Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre
Locations (1):
- Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre, Hyderabad, Andhra Pradesh, India